CLINICAL TRIAL: NCT00160173
Title: Efficacy Study Comparing 0.9 g and 1.25 g EstroGelÂ® 0.03% Doses With Placebo in the Treatment of Vasomotor Symptoms and Vulvar and Vaginal Atrophy Associated With Menopause
Brief Title: Efficacy Study Comparing 0.9 g and 1.25 g Estrogel With Placebo for Vasomotor Symptoms and Vulvar and Vaginal Atrophy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ASCEND Therapeutics (Industry)
Collaborators: Solvay Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S166.4.003
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Postmenopausal Symptoms
Keywords: Post menopausal vasomotor symptoms
MeSH Terms: interventions — Estradiol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- EstroGel® Gel 0.9 grams 0.03% (Experimental): 0.9 g of EstroGel® 0.03% applied to one arm and 1.25 g of placebo gel applied on the other arm once daily for 12 weeks.
  Interventions: Drug: Estrogel
- EstroGel® Gel 1.25 grams 0.03% (Experimental): 1.25 g of EstroGel® 0.03% applied to one arm and 0.9 g of placebo gel applied on the other arm once daily for 12 weeks.
  Interventions: Drug: Estrogel
- Placebo Gel (Placebo Comparator): 0.9 g of placebo gel applied to one arm and 1.25 g of placebo gel applied on the other arm once daily for 12 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Estrogel
  Arms: EstroGel® Gel 0.9 grams 0.03%; EstroGel® Gel 1.25 grams 0.03%
Other: Placebo
  Arms: Placebo Gel

SUMMARY:
This study is intended to establish the lowest effective dose of EstroGel® for the treatment of vasomotor symptoms associated with menopause.

DETAILED DESCRIPTION:
The primary objective of this study was to establish the lowest effective dose of EstroGel® for the treatment of vasomotor symptoms associated with menopause by comparing the efficacy of 0.9 g and 1.25 g EstroGel® 0.03% doses with placebo. Effects on symptoms of vulvar and vaginal atrophy were assessed as secondary efficacy parameters.

ELIGIBILITY:
Inclusion Criteria:

* Women 45-65 years
* naturally or surgically postmenopausal
* experiencing hot flushes

Exclusion Criteria:

* hypersensitivity to estrogen replacement therapy
* pregnancy or lactating
* abnormal PAP smear
* history/suspected cervical, uterine, adrenal, pituitary, breast or ovarian malignancy

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2004-12-02 (Actual); Primary Completion 2005-09-06 (Actual); Study Completion 2005-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (109):
- United States (109):
  - Site 112, Birmingham, Alabama
  - Site 74, Mobile, Alabama
  - Site 20, Montgomery, Alabama
  - Site 34, Tucson, Arizona
  - Site 68, Tucson, Arizona
  - Site 5, Jonesboro, Arkansas
  - Site 88, Little Rock, Arkansas
  - Site 95, Little Rock, Arkansas
  - Site 104, Carmichael, California
  - Site 42, Encinitas, California
  - Site 21, San Diego, California
  - Site 37, San Diego, California
  - Site 78, San Diego, California
  - Site 82, San Diego, California
  - Site 69, Avon, Connecticut
  - Site 58, Bridgeport, Connecticut
  - Site 3, Groton, Connecticut
  - Site 72, Hartford, Connecticut
  - Site 54, New Britain, Connecticut
  - Site 79, Southport, Connecticut
  - Site 18, Waterbury, Connecticut
  - Site 97, West Hartford, Connecticut
  - Site 35, Aventura, Florida
  - Site 36, Aventura, Florida
  - Site 105, Clearwater, Florida
  - Site 49, Clearwater, Florida
  - Site 91, Daytona Beach, Florida
  - Site 57, Melbourne, Florida
  - Site 109, Miami, Florida
  - Site 39, Pinellas Park, Florida
  - Site 107, Spring Hill, Florida
  - Site 100, Tampa, Florida
  - Site 77, West Palm Beach, Florida
  - Site 61, Alpharetta, Georgia
  - Site 81, Alpharetta, Georgia
  - Site 28, Atlanta, Georgia
  - Site 93, Atlanta, Georgia
  - Site 55, Decatur, Georgia
  - Site 13, Douglasville, Georgia
  - Site 87, Powder Springs, Georgia
  - Site 22, Savannah, Georgia
  - Site 99, Savannah, Georgia
  - Site 53, Boise, Idaho
  - Site 96, Champaign, Illinois
  - Site 24, Chicago, Illinois
  - Site 84, Chicago, Illinois
  - Site 26, Peoria, Illinois
  - Site 46, Peoria, Illinois
  - Site 75, Evansville, Indiana
  - Site 45, South Bend, Indiana
  - Site 8, Waterloo, Iowa
  - Site 108, Lexington, Kentucky
  - Site 50, Baton Rouge, Louisiana
  - Site 12, Metairie, Louisiana
  - Site 65, New Orleans, Louisiana
  - Site 16, Shreveport, Louisiana
  - Site 11, Baltimore, Maryland
  - Site 66, Ann Arbor, Michigan
  - Site 15, Chaska, Minnesota
  - Site 29, Creve Coeur, Missouri
  - Site 2, St Louis, Missouri
  - Site 67, St Louis, Missouri
  - Site 19, Billings, Montana
  - Site 56, Lincoln, Nebraska
  - Site 6, Las Vegas, Nevada
  - Site 40, Reno, Nevada
  - Site102, Olean, New York
  - Site 31, Fayetteville, North Carolina
  - Site 60, New Bern, North Carolina
  - Site 59, Raleigh, North Carolina
  - Site 38, Winston-Salem, North Carolina
  - Site 70, Winston-Salem, North Carolina
  - Site 85, Winston-Salem, North Carolina
  - Site 86, Cincinnati, Ohio
  - Site 101, Edmond, Oklahoma
  - Site 89, Eugene, Oregon
  - Site 111, Medford, Oregon
  - Site 64, Portland, Oregon
  - Site 113, Erie, Pennsylvania
  - Site 98, Pottstown, Pennsylvania
  - Site 33, Greenville, South Carolina
  - Site 9, Chattanooga, Tennessee
  - Site 92, Memphis, Tennessee
  - Site 76, Nashville, Tennessee
  - Site 83, Carrollton, Texas
  - Site 17, Conroe, Texas
  - Site 23, Corpus Christi, Texas
  - Site 25, Corpus Christi, Texas
  - Site 30, Dallas, Texas
  - Site 90, Dallas, Texas
  - Site 10, Houston, Texas
  - Site 110, Houston, Texas
  - Site 14, Houston, Texas
  - Site 27, Houston, Texas
  - Site 48, Houston, Texas
  - Site 51, Houston, Texas
  - Site 71, Houston, Texas
  - Site 73, Houston, Texas
  - Site 43, San Antonio, Texas
  - Site 62, San Antonio, Texas
  - Site 80, San Antonio, Texas
  - Site 7, Texarkana, Texas
  - Site 44, Salt Lake City, Utah
  - Site 94, Salt Lake City, Utah
  - Site 47, Norfolk, Virginia
  - Site 106, Richmond, Virginia
  - Site 41, Richmond, Virginia
  - Site 4, Seattle, Washington
  - Site 52, Tacoma, Washington